CLINICAL TRIAL: NCT05237349
Title: A Prospective, Single-arm Clinical Trial of Envafolimab Combined With Chemotherapy in Metastatic or Recurrent Gastric Adenocarcinoma
Brief Title: Envafolimab Combined With Chemotherapy in Metastatic or Recurrent Gastric Adenocarcinoma
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Liangjun Zhu M.M. (Other)
Collaborators: Zhangjiagang First People's Hospital (Other)
Responsible Party: Sponsor-Investigator, Liangjun Zhu M.M., chief physician, Jiangsu Cancer Institute & Hospital
Organization: Jiangsu Cancer Institute & Hospital (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: SMA-GC-001
Record Dates: First submitted 2022-01-18; First posted 2022-02-14 (Actual); Last update posted 2024-01-05 (Actual); Status verified 2024-01

CONDITIONS: Metastatic or Recurrent Gastric Adenocarcinoma
MeSH Terms: conditions — Neoplasm Metastasis | interventions — envafolimab; Immunotherapy; Oxaliplatin; Drug Therapy; S 1 (combination)

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- envafolimab plus chemotherapy (Experimental): Envafolimab:300mg,sc,d1,Q3W; Chemotherapy:SOX(Oxaliplatin，130mg/m2, iv,d1,Q3W + S-1，40mg/m2, op,bid,d1-14,Q3W).
  Interventions: Drug: Envafolimab; Drug: Oxaliplatin; Drug: S1

INTERVENTIONS:
Drug: Envafolimab — 300mg,sc,d1,Q3W
  Other Names: Immunotherapy
Drug: Oxaliplatin — 130mg/m2, iv,d1,Q3W
  Other Names: Chemotherapy
Drug: S1 — 40mg/m2, op,bid,d1-14,Q3W
  Other Names: Chemotherapy

SUMMARY:
The objective is to investigate the efficacy and safety of Envafolimab combined with chemotherapy in the treatment of metastatic or recurrent gastric adenocarcinoma.

DETAILED DESCRIPTION:
Envafolimab indication: Envafolimab is the world's first subcutaneous injection of PD-L1 monoclonal antibody.Suitable for adult patients with advanced solid tumors with unresectable or metastatic microsatellite highly unstable (MSI-H) or mismatch repair gene defects (dMMR).

ELIGIBILITY:
Inclusion Criteria:

* 18-75 years；
* ECOG 0-1；
* life expectancy of at least 3 months；
* Negative for HER2 gene expression by central laboratory ；
* The tumor expresses PD-L1 as detected by the central laboratory, and the tumor proportion score (CPS) ≥ 1；
* At least one measurable objective tumor lesion by spiral CT examination, the maximum diameter ≥ 1cm（according to RECIST 1.1）；
* Diagnosed by histology and/or cytology, and assessed by imaging (refer to RECIST 1.1) as advanced metastatic gastric adenocarcinoma or gastric adenocarcinoma that has recurred after previous gastric cancer surgery;
* Not received systemic chemotherapy in the past. Patients who have previously received fluorouracil monotherapy or fluorouracil-based adjuvant therapy or neoadjuvant therapy, and patients who have completed adjuvant therapy or neoadjuvant therapy before the start of the chemotherapy regimen in this trial 6 months ago can be included in this trial. In cases of metastatic disease requiring local remission, remission therapy with radiosensitizing doses of fluorouracil or capecitabine alone is permitted only ；
* satisfactory main organ function，laboratory test must meet the following criteria: hemoglobin (HGB) ≥90g/L, neutrophil count（ANC） ≥1.5×109/L, platelet count（PLT） ≥80×109/L, Serum creatinine（CR）≤1.5 upper normal limitation (UNL)，total bilirubin (TBil) ≤1.5 upper normal limitation (UNL), alanine aminotransferase (ALT) and aspartate aminotransferase (AST) ≤2.5 UNL (For patients with liver metastasis, the AST/ALT must be ≤5.0 UNL), Activated partial thromboplastin time (APTT), international normalized ratio (INR), prothrombin time (PT) ≤ 1.5×ULN; left ventricular ejection fraction (LVEF) ≥ 50%; thyroid stimulating hormone (TSH) within the normal range Within: if the baseline TSH exceeds the normal range, subjects with total T3 (or FT3) and FT4 within the normal range can also be enrolled;
* Subjects of childbearing potential must use an appropriate method of contraception during the study period and within 120 days after the end of the study, have a negative serum pregnancy test within 7 days prior to study enrollment, and must be non-lactating subjects ；

Exclusion Criteria:

* Suffered from other malignant tumors within 5 years before the start of treatment in this study;
* Pathologically suggested patients with abnormally increased AFP OR MSI-H ；
* Grade ≥1 unresolved toxicities (according to the most recent version of the National Cancer Institute [NCI] Common Terminology Criteria for Adverse Events [CTCAE]) due to any prior therapy, excluding alopecia and fatigue; neurotoxicity was Recovery to ≤ grade 1 or baseline before the group;
* Subjects with any severe and/or uncontrolled disease ；
* Poorly controlled diabetes (fasting blood glucose [FBG] > 10 mmol/L) ；
* Received major surgical treatment, incisional biopsy, or significant traumatic injury within 28 days prior to the start of study treatment; or had a long-term unhealed wound or fracture；
* Serious arterial/venous thrombotic event within 6 months prior to initiation of study treatment ；
* Previously received drug therapy against PD-1, PD-L1 and other related immune checkpoints ；
* Participating in or participating in other clinical investigators within 4 weeks prior to the start of the study ；
* Allergic to the active ingredients or excipients of the study drug ；
* Unsuitable for the study or other chemotherapy determined by investigator.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2024-12-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
ORR | 6 months
  Objective response rate

SECONDARY OUTCOMES:
PFS | 6 months
  Progression Free Survival
OS | 12 months
  Overall Survival
DCR | 9 months
  Disease Control Rate
DOR | 12 months
  Duration of Response
AEs | 12 months
  Percentage of participants experiencing grade 3-5 adverse events
Qualify of Life | 12 months
  Based on Quality of Life Questionnare-Core 30, evaluate the quality of life of patients

CONTACTS AND LOCATIONS:
Overall Officials: Liangjun Zhu, Study Chair — Jiangsu Cancer Institute & Hospital
Locations (1):
- Jiangsu Cancer Institute & Hospital, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No